CLINICAL TRIAL: NCT02530463
Title: Combination of Nivolumab and Ipilimumab With 5-Azacitidine in Patients With Myelodysplastic Syndromes (MDS)
Brief Title: Nivolumab and/or Ipilimumab With or Without Azacitidine in Treating Patients With Myelodysplastic Syndrome
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0930; NCI-2015-01494 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0930 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-08-19; First posted 2015-08-21 (Estimated); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Leukemia; Myelodysplastic Syndrome; Recurrent Myelodysplastic Syndrome
Keywords: Leukemia; Myelodysplastic syndrome; MDS; Nivolumab; BMS-936558; Opdivo; Ipilimumab; Yervoy; BMS-734016; MDX010; 5-azacitidine; Azacitidine; 5-AZA; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816; Azacytidine
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes | interventions — Azacitidine; Ipilimumab; CTLA-4 Antigen; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort I (nivolumab) (Experimental): Patients receive nivolumab IV over 30 minutes on days 1 and 15. Treatment repeats every 4 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients with disease progression may receive nivolumab and azacitidine at the discretion of the treating physician.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Nivolumab
- Cohort II (ipilimumab) (Experimental): Patients receive ipilimumab IV over 30 minutes on day 1. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients with disease progression may receive ipilimumab and azacitidine at the discretion of the treating physician.
  Interventions: Biological: Ipilimumab; Other: Laboratory Biomarker Analysis
- Cohort III (nivolumab, ipilimumab) (Experimental): Patients receive nivolumab IV over 30 minutes on days 1 and 15 and ipilimumab IV over 30 minutes on day 1. Treatment repeats every 4 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive nivolumab IV over 30 minutes every 2 weeks (or every 4 weeks if patients receive azacitidine) in the absence of disease progression or unacceptable toxicity. Patients with disease progression may receive ipilimumab, nivolumab, and azacitidine at the discretion of the treating physician.
  Interventions: Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Biological: Nivolumab
- Cohort IV (azacitidine, nivolumab) (Experimental): Patients receive azacitidine IV over 10-40 minutes on days 1-5 and nivolumab IV over 30 minutes on days 6 and 20. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Other: Laboratory Biomarker Analysis; Biological: Nivolumab
- Cohort V (azacitidine, ipilimumab) (Experimental): Patients receive azacitidine IV over 10-40 minutes on days 1-5 and ipilimumab IV over 30 minutes on day 6. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Biological: Ipilimumab; Other: Laboratory Biomarker Analysis
- Cohort VI (azacitidine, nivolumab, ipilimumab) (Experimental): Patients receive azacitidine IV over 10-40 minutes on days 1-5 and nivolumab IV over 30 minutes and ipilimumab IV over 30 minutes on day 6. Treatment with ipilimumab repeats every 4 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Cycles with nivolumab and azacitidine repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Biological: Nivolumab

INTERVENTIONS:
Drug: Azacitidine — Given IV
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
  Arms: Cohort IV (azacitidine, nivolumab); Cohort V (azacitidine, ipilimumab); Cohort VI (azacitidine, nivolumab, ipilimumab)
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
  Arms: Cohort II (ipilimumab); Cohort III (nivolumab, ipilimumab); Cohort V (azacitidine, ipilimumab); Cohort VI (azacitidine, nivolumab, ipilimumab)
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
  Arms: Cohort I (nivolumab); Cohort III (nivolumab, ipilimumab); Cohort IV (azacitidine, nivolumab); Cohort VI (azacitidine, nivolumab, ipilimumab)

SUMMARY:
This phase II trial studies the side effects of nivolumab and/or ipilimumab with or without azacitidine and to see how well they work in treating patients with myelodysplastic syndrome. Monoclonal antibodies, such as nivolumab and ipilimumab, may block cancer growth in different ways by targeting certain cells. Drugs used in chemotherapy, such as azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving nivolumab and/or ipilimumab with or without azacitidine may work better in treating myelodysplastic syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of nivolumab and ipilimumab, as single agents or in combination and with 5-azacitidine (azacitidine), in patients with myelodysplastic syndrome (MDS).

SECONDARY OBJECTIVES:

I. To explore the clinical activity of nivolumab and ipilimumab, as single agents or in combination and with 5-azacitidine, in patients with MDS.

II. To explore the biological activity of these compounds in patients with MDS.

OUTLINE: Patients are assigned to 1 of 6 cohorts. Patients with hypomethylating failure MDS are assigned to cohorts I, II, or III. Patients with previously untreated MDS are assigned to cohorts IV, V, or VI.

COHORT I (COHORT COMPLETED AS OF 10/7/19): Patients receive nivolumab intravenously (IV) over 30 minutes on days 1 and 15. Treatment repeats every 4 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients with disease progression may receive nivolumab and azacitidine at the discretion of the treating physician.

COHORT II (COHORT COMPLETED AS OF 10/7/19): Patients receive ipilimumab IV over 30 minutes on day 1. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients with disease progression may receive ipilimumab and azacitidine at the discretion of the treating physician.

COHORT III: Patients receive nivolumab IV over 30 minutes on days 1 and 15 and ipilimumab IV over 30 minutes on day 1. Treatment repeats every 4 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive nivolumab IV over 30 minutes every 2 weeks (or every 4 weeks if patients receive azacitidine) in the absence of disease progression or unacceptable toxicity. Patients with disease progression may receive ipilimumab, nivolumab, and azacitidine at the discretion of the treating physician.

COHORT IV (COHORT COMPLETED AS OF 10/7/19): Patients receive azacitidine IV over 10-40 minutes on days 1-5 and nivolumab IV over 30 minutes on days 6 and 20. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

COHORT V: Patients receive azacitidine IV over 10-40 minutes on days 1-5 and ipilimumab IV over 30 minutes on day 6. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

COHORT VI (COHORT ON-HOLD AS OF 10/7/19): Patients receive azacitidine IV over 10-40 minutes on days 1-5 and nivolumab IV over 30 minutes and ipilimumab IV over 30 minutes on day 6. Treatment with ipilimumab repeats every 4 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Cycles with nivolumab and azacitidine repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with MDS (up to 20% blasts) of any risk as defined as:

  * Previously untreated
  * Previously treated with hypomethylating agent (HMA) agent; patients need to have relapsed or progressed after any number of cycles of HMA therapy; patients that do not respond to HMA therapy will also be allowed in the study; relapse or progression will be measured by International Working Group (IWG) 2006 criteria; no response will be lack of clinical benefit after at least 6 cycles of HMA therapy
* Creatinine =< 2.0 x upper limit of normal (ULN)
* Serum bilirubin =< 2.0 x ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.0 x ULN
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Females of childbearing potential must have a negative serum or urine beta human chorionic gonadotropin (beta-hCG) pregnancy test result within 24 hours prior to the first dose of treatment and must agree to use an effective contraception method to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drugs; females of non-childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy
* Males who have partners of childbearing potential must agree to use an effective contraceptive method during the study and a period of 31 weeks after the last dose of investigational drug
* Patients or their legally authorized representative must provide written informed consent

Exclusion Criteria:

* Second malignancy currently requiring active therapy, except breast or prostate cancer stable on or responding to endocrine therapy
* Any major surgery, radiotherapy, chemotherapy, biologic therapy, immunotherapy, experimental therapy within 2 weeks prior to the first dose of the study drugs
* Patients with any other known concurrent severe and/or uncontrolled medical condition (e.g. uncontrolled diabetes; cardiovascular disease including congestive heart failure New York Heart Association [NYHA] class III or IV, myocardial infarction within 6 months, and poorly controlled hypertension; chronic renal failure; or active uncontrolled infection) which, in the opinion of the investigator could compromise participation in the study
* Patients unwilling or unable to comply with the protocol
* History of pneumonitis
* Patients who are on high dose steroid (equivalent of prednisone more than 10 mg a day) or immune suppression medications
* Patients with autoimmune diseases (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's granulomatosis])
* Patients with a history of inflammatory bowel disease such as Crohn's disease and ulcerative colitis
* Patients known to be positive for hepatitis B surface antigen expression or with active hepatitis C infection (positive by polymerase chain reaction or on antiviral therapy for hepatitis C within the last 6 months); patients with history of human immunodeficiency virus (HIV) disease are also excluded from the study
* Current therapy with other systemic anti-neoplastic or anti-neoplastic investigational agents
* Females who are pregnant or lactating
* Prior treatment with allogeneic stem cell transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2015-09-08 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) in MDS Participants with Hypomethylating Agent Failure | 24 weeks
  Overall response rate (ORR) defined as complete response plus partial response (CR + PR) + hematological improvement (HI).
Overall Response Rate (ORR) in MDS Participants Who Have Not Received Hypomethylating Agents | 30 weeks
  Overall response rate (ORR) defined as complete response plus partial response (CR + PR) + hematological improvement (HI).

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Garcia-Manero, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org